CLINICAL TRIAL: NCT06898307
Title: Utility of Gene Test Analysis for Diagnosis, Prognosis and Treatment of Patients With Genetic Arrhythmic Heart Disease: the ARRHYTHMIC GENE-HEART
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Other Study IDs: 307/2023/Oss/AOUFe
Record Dates: First submitted 2025-03-03; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Genetic Disease; Cardiac Disease; Cardiac Arrhythmias; Genetic Disorder; Cardiology
Keywords: Cardiogenetic
MeSH Terms: conditions — Genetic Diseases, Inborn; Heart Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cardiogenetic disease

SUMMARY:
The goal of this observational study is to enroll all patients evaluated at the specialized Cardiogenetic Center within the Cardiology Department of the University of Ferrara, Italy. The primary aim of the registry is to collect comprehensive clinical, genetic, and electrophysiological data from individuals with suspected or confirmed arrhythmogenic conditions. By systematically documenting patient demographics, family history, clinical presentations, diagnostic findings, and treatment outcomes, the registry seeks to enhance our understanding of the genetic basis and clinical implications of genetically driven arrhythmias and systemic syndromes. This registry will facilitate long-term follow-up of enrolled patients to assess the natural history of arrhythmogenic disorders and the effectiveness of various therapeutic interventions. Additionally, it aims to identify potential risk factors associated with adverse outcomes, such as sudden cardiac death or major arrhythmic events.

DETAILED DESCRIPTION:
Cardiogenetics is essential in daily clinical practice, providing critical insights into the genetic basis of inherited cardiovascular conditions. This knowledge enables more accurate diagnoses, risk assessments, and personalized management strategies for patients. By understanding the genetic underpinnings of arrhythmias and other heart diseases, healthcare providers can identify at-risk individuals and their family members, facilitating early intervention and preventive measures. Establishing an observational registry for these conditions is vital, as it systematically collects data on patient demographics, clinical presentations, genetic findings, and treatment outcomes. This comprehensive database enhances our understanding of the natural history and variability of genetic cardiovascular disorders while supporting research efforts aimed at developing improved diagnostic tools and therapeutic approaches. Ultimately, such a registry can enhance patient care by informing clinical guidelines and fostering collaboration among clinicians, geneticists, and researchers in the field.

Therefore, the goal of this observational study is to gather extensive clinical, genetic, and electrophysiological data from individuals with suspected or confirmed arrhythmogenic conditions. By systematically documenting patient demographics, family history, clinical presentations, diagnostic findings, and treatment outcomes, the registry aims to deepen our understanding of the genetic basis and clinical implications of genetically driven arrhythmias and systemic syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated at the Cardiogenetic Center of the University of Ferrara in Ferrara, Italy.
* Having a proven cardiogenetic disease

Exclusion Criteria:

* Refuse to provide informed consents
* Patients not having a cardiogenic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
All-cause of death | At one and 5 years (end of the study)
  The investigators will monitor patient's all causes death
Cardiovascular-related death | At one and 5 years (end of the study)
  The investigators will monitor patient's all causes death

SECONDARY OUTCOMES:
Onset or worsening heart faillure | At one and 5 years (end of the study)
  The investigators will assess patient's hemodynamic stability over the years, monitoring the onset or the worsening of heart failure
Onset/worsening of atrial tachyarrhythmias | At one and 5 years (end of the study)
Onset/worsening of ventricular tachyarrhythmias | At one and 5 years (end of the study)
  The investigators will monitor patient's rhythm over the years, assessing the onset or the worsening of ventricular tachyarrhythmias.
Need for PM/ICD | At one and 5 years (end of the study)
  The investigators will evaluate procedural time of different cardiac pacing modalities
Types of genetic mutations | At the time of genetic analysis
  Types of genetic mutations

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Balla, MD PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Department of Cardiology, University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conte G, Wilde A, Behr ER, Scherr D, Lenarczyk R, Gandjbachkh E, Crotti L, Brugada-Sarquella G, Potpara T. Importance of Dedicated Units for the Management of Patients With Inherited Arrhythmia Syndromes. Circ Genom Precis Med. 2021 Apr;14(2):e003313. doi: 10.1161/CIRCGEN.120.003313. Epub 2021 Apr 2. No abstract available. PMID 33797288
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Background] Wilde AA, Behr ER. Genetic testing for inherited cardiac disease. Nat Rev Cardiol. 2013 Oct;10(10):571-83. doi: 10.1038/nrcardio.2013.108. Epub 2013 Jul 30. PMID 23900354
- [Background] Priori SG, Wilde AA, Horie M, Cho Y, Behr ER, Berul C, Blom N, Brugada J, Chiang CE, Huikuri H, Kannankeril P, Krahn A, Leenhardt A, Moss A, Schwartz PJ, Shimizu W, Tomaselli G, Tracy C. HRS/EHRA/APHRS expert consensus statement on the diagnosis and management of patients with inherited primary arrhythmia syndromes: document endorsed by HRS, EHRA, and APHRS in May 2013 and by ACCF, AHA, PACES, and AEPC in June 2013. Heart Rhythm. 2013 Dec;10(12):1932-63. doi: 10.1016/j.hrthm.2013.05.014. Epub 2013 Aug 30. No abstract available. PMID 24011539